CLINICAL TRIAL: NCT06069856
Title: Individually Randomized Crossover Trial of Multiple Micronutrient Supplementation (MMS) Versus IFA During Pregnancy in Tanzania
Brief Title: Multiple Micronutrient Supplementation (MMS) vs IFA Acceptability Crossover Trial
Acronym: MIFA-ACT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Ifakara Health Institute (Other); Harvard School of Public Health (HSPH) (Other); Muhimbili University of Health and Allied Sciences (Other); Africa Academy for Public Health (Other); Columbia University (Other)
Responsible Party: Principal Investigator, Emily Smith, Principal Investigator, George Washington University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: MIFA-ACT
Record Dates: First submitted 2023-09-15; First posted 2023-10-06 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Pregnancy Related
Keywords: Acceptability; Multiple Micronutrient Supplementation; Iron; IFA; Tanzania
MeSH Terms: interventions — Iron

STUDY DESIGN:
Masking Description: None (Open label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MMS with 60 mg of iron first, then IFA with 60 mg of iron (Experimental): Women will receive the first regimen (MMS with 60 mg of iron) for 2 months and then crossover on to the second regimen (IFA with 60 mg of iron) for 2 months
  Interventions: Dietary Supplement: Iron Folic Acid Tablets with 60 mg of iron; Dietary Supplement: Multiple Micronutrient Supplements with 60 mg of elemental iron
- IFA with 60 mg of iron first, then MMS with 60 mg of iron (Experimental): Women will receive the first regimen (IFA with 60 mg of iron) for 2 months and then crossover on to the second regimen (MMS with 60 mg of iron) for 2 months
  Interventions: Dietary Supplement: Iron Folic Acid Tablets with 60 mg of iron; Dietary Supplement: Multiple Micronutrient Supplements with 60 mg of elemental iron

INTERVENTIONS:
Dietary Supplement: Iron Folic Acid Tablets with 60 mg of iron — IFA with 60 mg iron is an intervention group. IFA with 60 mg of iron will be taken orally once daily from the time of randomization
Dietary Supplement: Multiple Micronutrient Supplements with 60 mg of elemental iron — MMS with 60 mg iron is an intervention group. MMS with 60 mg of iron plus standard UNIMMAP formulation for other 14 micronutrients will be taken orally once daily from the time of randomization.

SUMMARY:
This is an open-label individually randomized mixed methods cross-over trial to assess acceptability, preference, and side effects of IFA formulations with 60 mg of iron to MMS formulations with 60 mg of iron.

ELIGIBILITY:
Inclusion Criteria:

* Attending first ANC visit at the study clinic
* Pregnant women ≤ 15 weeks of gestation
* Aged ≥ 18 years
* Intending to stay in the study area for the duration of study
* Provides informed consent

Exclusion Criteria:

* Severe anemia (defined as Hb <8.5 g/dL per Tanzania standard of care)
* Sickle cell disease (SS,SC, CC genotype) as tested by HemoTypeSC
* Concurrent participation in other nutritional supplementation trial
* Pregnant women with disability or condition which would impair their ability to provide informed consent and complete study procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Acceptability of formulation | At two months of taking each regimen
  To assess acceptability of MMS formulation with 60 mg of iron and IFA formulation with 60 mg of iron using Likert scales ranging from 1 (disliked a lot) to 5 (liked a lot).

SECONDARY OUTCOMES:
Most preferred formulation | At four months (after taking both regimens)
  To assess participated reported preference of MMS formulation with 60 mg of iron and IFA formulation with 60 mg of iron by asking participants which supplement they like the best.
Side Effects of formulation | At two months of taking each regimen
  To assess the percentage of patients experiencing side effects of MMS formulation with 60 mg of iron and IFA formulation with 60 mg of iron
Adherence | At two months of taking each regimen
  Percentage pill count of the number of supplements taken

CONTACTS AND LOCATIONS:
Overall Officials: Blair Wylie, MD, MPH, Principal Investigator — Columbia University; Honorati Masanja, PhD, Principal Investigator — Ifakara Health Institute; Alfa Muhihi, PhD, Principal Investigator — Africa Academy of Public Health; Andrea Pembe, MD, MMed, PhD, FCOG, Principal Investigator — Muhimbili University of Health and Allied Sciences; Emily R Smith, ScD, MPH, Principal Investigator — The George Washington University; Christopher R Sudfeld, ScD, ScM, Principal Investigator — Harvard University